CLINICAL TRIAL: NCT00270790
Title: A SINGLE SITE EVALUATION OF AMIFOSTINE FOR MUCOSAL AND HEMOPOETIC PROTECTION AND CONCURRENT CARBOPLATIN, TAXOL, RADIOTHERAPY IN THE MANAGEMENT OF PATIENTS WITH ADVANCED LOCOREGIONAL SQUAMOUS CELL CARCINOMAS OF THE HEAD AND NECK.
Brief Title: EVALUATION OF AMIFOSTINE FOR MUCOSAL AND HEMOPOETIC PROTECTION AND CARBOPLATIN, TAXOL, RADIOTHERAPY IN THE MANAGEMENT OF PATIENTS WITH HEAD AND NECK CANCER.(GCC 0202)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mohan Suntharalingam (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor-Investigator, Mohan Suntharalingam, Principal Investigator, University of Maryland
Organization: University of Maryland, Baltimore (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00021746
Record Dates: First submitted 2005-12-23; First posted 2005-12-28 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Amifostine; Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMIFOSTINE +CARBOPLATIN, TAXOL +RT (Experimental): EVALUATION OF AMIFOSTINE FOR MUCOSAL AND HEMOPOETIC PROTECTION AND CARBOPLATIN, TAXOL, RADIOTHERAPY IN THE MANAGEMENT OF PATIENTS WITH HEAD AND NECK CANCER.
  Interventions: Drug: Amifostine; Drug: Carboplatin; Drug: Taxol; Device: Radiotherapy

INTERVENTIONS:
Drug: Amifostine — Amifostine will be given at dose of 500 mg IV within one hour before radiation
Drug: Carboplatin — Carboplatin for 100 mg/m2 and will be administered after the taxol infusion
Drug: Taxol — Taxol will be given at a dose of 40 mg/m2 as a 3 hour infusion dose
Device: Radiotherapy — Radiation will be given at a dose of 1.8 Gy. for a total of 70.2 Gy

SUMMARY:
Purpose of this study:

There is some evidence that the best treatment for head and neck cancer involves a combination of radiation therapy and chemotherapy. Radiation therapy is a form of cancer treatment using high energy x-rays. Chemotherapy is a form of cancer treatment that uses special medications. This study uses two chemotherapy drugs (Taxol and Carboplatin), which are FDA approved for treating head and neck cancers. This treatment combination has been associated with difficulty, pain, or a burning sensation upon swallowing (called esophagitis), and decrease in blood cells (cells in the blood which fight against infection). The purpose of this study is to investigate whether the addition of another drug, Amifostine, can reduce the side effects of current combination treatment (radiation and chemotherapy which is standard of care). The addition of Amifostine is the investigational part of the study. The research study is also looking at the side effects of Amifostine and cancer's growth response to this combination treatment.

DETAILED DESCRIPTION:
Patients presenting with locally advanced squamous cell carcinomas of head and neck (SCCHN) continue to represent a significant therapeutic challenge. The bulk of tumor burden often proves to be overwhelming for conventional radiotherapy. Attempts to improve upon these poor outcomes have led investigators to explore several new strategies, one such being chemoradiation. One of the trials conducted at the University of Maryland with carboplatin and paclitaxel with daily radiation showed 82% CR at the primary site. But the most commonly encountered grade 3 toxicities were mucositis (70%), leukopenia (30%) and 3% grade 4 leukopenia. Amifostine: An organic thiophosphate is radioprotective and has shown to protect experimental animals from lethal doses of radiation. Clinical trials have demonstrated that amifostine can provide protection against the hematological toxicities and mucositis seen with various chemotherapeutic agents. Theoretically, drug interactions between amifostine and chemotherapeutic agents are not likely to occur, due to amifostine¿s rapid clearance from plasma (90% of the drug is cleared within 6 minutes). A promising venue would be the investigation of amifostine¿s role in reducing the toxicities associated with chemoradiation (which is standard of care of treating squamous cell carcinomas of head and neck).

Principal objectives of the study: Primary: To evaluate whether the addition of the radioprotector amifostine can reduce the incidence and severity of mucositis and hematological toxicities caused by chemoradiation. Secondary: 1.To determine the toxicities of amifostine given in this setting. 2. To determine the response rate of this regimen in the population.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proved locally advanced squamous cell carcinoma of the head and neck of all primary sites. The following TNM stages by sites will be eligible.

   Oral cavity, Pharynx, Larynx, Nasopharynx, paranasal sinuses: T4 N0-3, A,B,C T3 N1-3 A,B,C any T, N3 A,B,C Unknown primary: Tx, N3 A,B,C Note: Only clearly unresectable T4 N0 lesions are eligible for study provided the reasons for unresectability are due to extensive anatomic involvement and are outlined by the surgeon.
2. Karnofsky performance status of 70% or better at screen and on first day of treatment.
3. Patients with loco-regional recurrences from any site with no prior radiation therapy and not amenable for salvage surgery are eligible for study.
4. No evidence of distant metastatic disease.
5. No previous radiation therapy
6. No previous chemotherapy.
7. Adequate renal & bone marrow function determined by the following laboratory parameters.

   WBC 3500/ul or higher Platelet count 100.000/ul or higher Hemoglobin 9.0 g/dl or higher BUN 25 mg/dl or less, and Screatinine 2.0 mg/dl or less Total bilirubin less than 2.0 mg/dl, AST/ALT less than 3 times the ULN Creatinine Clearance 50 cc/min or higher
8. Evidence of measurable disease.
9. No evidence of concomitant malignancy except for non-melanomatous skin cancer (controlled or controllable) or carcinoma in situ of the cervix.
10. Signed informed consent.
11. No concomitant life threatening or uncontrolled serious medical illness such as end stage congestive heart failure cardiac arrythmia, liver disease and organic brain syndrome.
12. Age 18 years or older.

Exclusion Criteria:

1. Preexisting clinically significant neuropathy.
2. Patients currently taking antiarrhythmic medications are excluded.
3. History of poorly-controlled hypertension, angina, arrhythmias, or a history within the past 6 months of myocardial infarction or acute congestive heart failure.
4. Requirement for concurrent use of pilocarpine.
5. Treatment with any investigational drugs within 4 weeks of study entry.
6. Pregnant or lactating females or females of child bearing potential not employing adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2002-05; Primary Completion 2005-12 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Suntharalingam, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AMIFOSTINE +2 Chemo Lines +RT: EVALUATION OF AMIFOSTINE FOR MUCOSAL AND HEMOPOETIC PROTECTION AND CARBOPLATIN, TAXOL, RADIOTHERAPY IN THE MANAGEMENT OF PATIENTS WITH HEAD AND NECK CANCER.
  Amifostine: Amifostine will be given at dose of 500 mg IV within one hour before radiation
  Carboplatin: Carboplatin for 100 mg/m2
  Taxol: Taxol will be given at a dose of 40 mg/m2 as a 3 hour infusion dose
  Radiotherapy: Radiation will be given at a dose of 1.8 Gy. for a total of 70.2 Gy
Period: Overall Study
Arm/Group | AMIFOSTINE +2 Chemo Lines +RT
Started | 21
Completed | 16
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- AMIFOSTINE +CARBOPLATIN, TAXOL +RT: EVALUATION OF AMIFOSTINE FOR MUCOSAL AND HEMOPOETIC PROTECTION AND CARBOPLATIN, TAXOL, RADIOTHERAPY IN THE MANAGEMENT OF PATIENTS WITH HEAD AND NECK CANCER.
  Amifostine: Amifostine will be given at dose of 500 mg IV within one hour before radiation
  Carboplatin: Carboplatin for 100 mg/m2
  Taxol: Taxol will be given at a dose of 40 mg/m2 as a 3 hour infusion dose
  Radiotherapy: Radiation will be given at a dose of 1.8 Gy. for a total of 70.2 Gy
Arm/Group | AMIFOSTINE +CARBOPLATIN, TAXOL +RT
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 58.2 [48 to 70]
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Participants With Mucositis and Hematological Toxicities With the Addition of Radioprotector Amifostine
Description: Blood work (CMP was collected and evaluated for neutropenia, leukopenia and anemia) is taken prior to chemotherapy administration. The toxicity levels were measured using Common Terminology Criteria for Adverse Events (CTCAE 3.0) and monitored based on the dose of Amifostine given.
Time Frame: 3 years
Population: 21 patients enrolled, however only 16 patients were analyzed due to 5 patients withdrawals.
Measure: Number; unit: participants
Arm/Group | AMIFOSTINE +CARBOPLATIN, TAXOL +RT
Number analyzed (Participants) | 16
participants | 16

2. Secondary Outcome: Response Rates Based on the Study Regimen
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 3 years
Population: 21 patients enrolled, however only 16 patients were analyzed due to 5 patients withdrawals.
Measure: Number; unit: participants
Arm/Group | AMIFOSTINE +CARBOPLATIN, TAXOL +RT
Number analyzed (Participants) | 16
participants | 16

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | AMIFOSTINE +CARBOPLATIN, TAXOL +RT
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 21/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMIFOSTINE +CARBOPLATIN, TAXOL +RT (N=21)
Fatigue (Investigations) | 21
Neutropenia (Blood and lymphatic system disorders) | 2
Mucositis (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 6
Xerostomia (Gastrointestinal disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Weight Loss (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No